CLINICAL TRIAL: NCT02279927
Title: Prospective Comparison Between Different Laser Settings for Ureteral \ Kidney Stones Treatment During
Brief Title: Prospective Comparison Between Different Laser Settings for Ureteral \ Kidney Stones Treatment During Ureteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMC-14-0063-CTIL
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Ureterolithiasis; Nephrolithiasis
Keywords: Ureteroscopy
MeSH Terms: conditions — Ureterolithiasis; Nephrolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low energy high frequency (Experimental): Ureteroscopy with laser settings of low energy & high frequency with aim of stone dusting
  Interventions: Device: Ureteroscopy
- High energy low frequency (Active Comparator): Ureteroscopy with laser settings of low energy high frequency with aim of stone fragmentation and basket extraction of fragments
  Interventions: Device: Ureteroscopy

INTERVENTIONS:
Device: Ureteroscopy — Ureteroscopy with laser stone fragmentation

SUMMARY:
A prospective study comparing different laser settings used for stone fragmentation during ureteroscopy

DETAILED DESCRIPTION:
Two groups prospectively randomized for different laser settings during ureteroscopy one aimed for stone dusting, the other for stone fragmentation and basket extraction of fragments

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for ureteroscopy \ retrograde intra renal surgery (RIRS) for stone treatment

Exclusion Criteria:

* known ureteral stricture
* severe immune deficiency
* patients after urinary diversion surgery
* patients with single \ ectopic\ implanted kidney
* double collecting system
* severe thrombocytopenia
* patients taking anticoagulant drugs that cannot be stooped before the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 1 month

SECONDARY OUTCOMES:
Duration of operation | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Freifeld, Principal Investigator — Carmel MC
Locations (1):
- Carmel Medical Center, Haifa, Israel